CLINICAL TRIAL: NCT06761534
Title: Development and Verification of a Screening Tool for Comprehensive Geriatric Assessment of Elderly Tumor Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, Director, Sichuan Cancer Hospital and Research Institute
Other Study IDs: EK2023004
Record Dates: First submitted 2024-12-28; First posted 2025-01-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Geriatric Assessment; Geriatric Patients; Patients With Cancer; Assessment Tool
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Elderly cancer patients: Elderly cancer patients were assessed with the screening tool and G8. If the patient's screening result is positive (frailty risk population), continue with the CGA.
  Interventions: Other: Screening of comprehensive geriatic assessment.; Other: the G8 assessment; Other: Comprehensive Geriatric Assessment (CGA)

INTERVENTIONS:
Other: Screening of comprehensive geriatic assessment. — The participants are screened before anti-tumor therapy with a comprehensive assessment screening tool developed for elderly cancer patients, which is more suitable for individualized decision-making in anti-tumor treatment.
Other: the G8 assessment — The G8 is a rapid geriatric screening test that takes only a few minutes to complete. It is used as a calibration standard to validate the novel screening tool in this study.
Other: Comprehensive Geriatric Assessment (CGA) — The participants screened as a high frailty risk will undergo CGA to determine the most appropriate treatment plan.

SUMMARY:
This study is an observational research.

1. The study first conducted an electronic questionnaire survey among clinicians working in general and specialized hospitals at various levels nationwide to understand the implementation status and influencing factors of comprehensive geriatric assessment (CGA) for elderly cancer patients in China.
2. Based on the survey results, an interview outline was developed, and semi-structured interviews were conducted with professional doctors experienced in the diagnosis and treatment of elderly cancer patients to further explore the comprehensive factors influencing the implementation of CGA for this population.
3. According to the feedback from the semi-structured interviews, the survey results, and literature reports, the assessment dimensions required for the CGA screening tool were selected. An expert consultation survey questionnaire was designed around these dimensions, and the most suitable assessment items under each dimension were determined using the Delphi expert consultation method.
4. The G8 scale was used to assess elderly cancer patients. Items were selected based on their performance to form the screening tool. By setting thresholds and allocating weights for each item, CGA Screening Tool 1.0 was developed.
5. Pre-testing and modification of the screening tool were conducted. Investigators used the initially formed screening tool to conduct one-on-one patient testing. Feedback on the tool's clarity, relevance, clinical applicability (localization), and feasibility was obtained through consultation with a clinical expert panel to improve and refine its content and management process. This led to the revision and formation of CGA Screening Tool 2.0.
6. The reliability and validity of the CGA screening tool were verified using classical measurement theory to ensure the stability, reliability, and effectiveness of the scale tool in practical applications.
7. Patients were assessed using both CGA and the screening tool. External validation of Screening Tool 2.0 was performed using CGA as the gold standard to further evaluate the sensitivity, specificity, and accuracy of the screening tool.
8. Patients who participated in the assessment during the study were followed up to compare the correlation between different assessment results and patient completion of anti-tumor treatment, treatment efficacy, and the risk of related adverse reactions. The impact of the CGA screening tool on the implementation of CGA and its predictive ability for anti-tumor treatment were explored. Study data were obtained from the electronic medical record database and hospital information system of Sichuan Cancer Hospital, including clinicopathological features such as gender, age, clinical stage at diagnosis, and information related to anti-tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old
2. There are clear pathological data to diagnose malignant tumors, and follow-up anti-tumor therapy is determined in this institution
3. Have a certain enthusiasm for this study, and voluntarily participate in this study

Exclusion Criteria:

1. Unable to understand the content of the research
2. Unable to cooperate with CGA and screening assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Among all participants, 316 were used to develop the screening tool, 10 for the pre-testing, and 132 for the reliability and validity testing of the screening scale. After the scale was completed, the remaining 220 patients were used for the external validation of the tool. Finally, all patients evaluated using the screening tool were grouped according to different screening results, and the treatment effects and risks among the groups were compared.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Baseline
  (Truly frail elderly patients assessed by the novel screening tool and G8) / (Truly frail risk patients + elderly patients with negative results from novel screening tool but actually at risk of frailty after G8 assessment

SECONDARY OUTCOMES:
Accuracy | Baseline
  (The number of elderly patients truly at risk of frailty assessed by the novel screening tool and G8 + the number of elderly patients truly without frailty risk) / Total number of elderly patients in the study
Specificity | Baseline
  (True elderly patients without frailty risk assessed by the novel screening tool and G8) / (True patients without frailty risk + elderly patients with positive results from novel screening tool but actually without frailty risk after G8 screening)

OTHER OUTCOMES:
ORR | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or the end of study, whichever came first, assessed up to 12 months.
  the sum percentage of participants with CR and PR assessed by RECIST v1.1 criteria every 8-12 weeks.
PFS | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months.
  Systemic Progression-Free Survival assessed by the investigators using RECIST V1.1.
AE | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months.
  Number and percentage of patents with treatment-related adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China